CLINICAL TRIAL: NCT01313377
Title: Phase III Multicenter Randomized Study Comparing the Effect of Adjuvant Chemotherapy for Six Months With Gemcitabine-Oxaliplatin 85 mg/m2 (GEMOX 85) to Observation in Patients Who Underwent Surgery for Cancer of the Bile Ducts
Brief Title: Gemcitabine Hydrochloride and Oxaliplatin or Observation in Treating Patients With Biliary Tract Cancer That Has Been Removed by Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000696193; FRE-FNCLCC-ACCORD-18/0803; FRE-FNCLCC-PRODIGE-12; EUDRACT-2008-004560-39; EU-20982
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Liver Cancer
Keywords: adenocarcinoma of the extrahepatic bile duct; cholangiocarcinoma of the extrahepatic bile duct; liver and intrahepatic biliary tract cancer; localized extrahepatic bile duct cancer; adenocarcinoma of the gallbladder; cholangiocarcinoma of the gallbladder; localized gallbladder cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Gemcitabine; Oxaliplatin; Watchful Waiting; Chemotherapy, Adjuvant

ARMS (2):
- ARM A: Gemox 85 (Experimental): Adjuvant chemotherapy for six months with gemcitabine - oxaliplatin 85mg / m² ( GEMOX 85)
  Interventions: Drug: gemcitabine hydrochloride; Drug: oxaliplatin; Procedure: adjuvant therapy; Procedure: quality-of-life assessment
- ARM B: (Other): Observation until progression or death
  Interventions: Other: clinical observation; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: gemcitabine hydrochloride
  Arms: ARM A: Gemox 85
Drug: oxaliplatin
  Arms: ARM A: Gemox 85
Other: clinical observation
  Arms: ARM B:
Procedure: adjuvant therapy
  Arms: ARM A: Gemox 85
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine hydrochloride and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Observation is watching a patient's condition but not giving treatment until symptoms appear. It is not yet known whether giving gemcitabine hydrochloride together with oxaliplatin is more effective than observation in treating patients with biliary tract cancer that has been removed by surgery.

PURPOSE: This randomized phase III trial is studying giving gemcitabine hydrochloride together with oxaliplatin to see how well it works compared with observation in treating patients with biliary tract cancer that has been removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare disease-free survival (DFS) of patients with resected biliary tract cancer treated with adjuvant gemcitabine hydrochloride and oxaliplatin versus clinical observation.
* Compare quality of life of these patients.

Secondary

* Compare overall survival of these patients.
* Determine the toxicity of the chemotherapy in these patients.
* Explore prognostic factors for DFS including resection result (R0 vs R1), location of primary tumor (intrahepatic vs extrahepatic vs gallbladder), evolution of CA19-9, and lymph node involvement (N0 vs N+ and Nx). (Exploratory)
* Study pathological factors in surgical specimens to identify main characteristics and phenotypic clinicoanatomical biliary tract cancers before therapy. (Exploratory)
* Identify nontumor-associated liver injury and factors that may facilitate the emergence of biliary tract cancers. (Exploratory)
* Identify signaling pathways that may predict response to therapy. (Exploratory)
* Determine the molecular characteristics to differentiate tumors according to their position in the biliary tract (extrahepatic bile duct, intrahepatic cholangiocarcinoma site [hilar], and peripheral cholangiocarcinoma vesicle site). (Exploratory)

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine hydrochloride IV over 100 minutes on day 1 and oxaliplatin IV over 2 hours on day 2. Treatment repeats every 14 days for 12 courses.
* Arm II: Patients undergo clinical observation only every 4 weeks for 5 months. Quality of life is assessed at baseline, at 3 and 6 months, and then at all follow-up visits.

After completion of study therapy, patients are followed up at 6 months, every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven adenocarcinoma of the intrahepatic bile ducts, gallbladder, or extrahepatic bile ducts

  * Mixed forms of hepatocholangiocarcinomas included provided the cholangiocarcinoma is predominant
* Underwent surgical resection of the disease (R0 or R1) at least 4 weeks but no more than 13 weeks ago
* Nonmetastatic disease as assessed by abdominal MRI and chest x-ray
* No cancer of the pancreas or duodenum invading the bile duct and ampulla of Vater

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Hemoglobin ≥ 10 g/dL (transfusion allowed)
* ANC ≥ 1,500/mm³
* Platelet count ≥ 75,000/mm³
* Creatinine clearance > 40 mL/min
* Prothrombin time > 60% OR INR < 1.5 (without anticoagulant therapy)
* Transaminases ≤ 5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Conjugated bilirubin ≤ 35 μmol/L (after biliary drainage, if necessary)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No contraindications to oxaliplatin and gemcitabine hydrochloride therapy
* Prior invasive cancer allowed provided it has been in complete remission for ≥ 5 years
* No other concurrent invasive cancer except adequately treated carcinoma in situ of the cervix or basal cell carcinoma
* No other severe, unresolved disease
* No mental illness
* No HIV positivity
* No grade 1 angina or symptomatic angina ≥ grade 2
* No sensitive peripheral neuropathy
* No uncontrolled diabetes
* No inability to undergo medical tests due to geographical, social, or psychological reasons
* No prisoners or patients under guardianship
* No Child B or C cirrhosis

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior neoadjuvant chemotherapy or radiotherapy
* No prior organ transplantation
* No concurrent participation in another clinical trial of an experimental agent

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2009-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | up to 3 years
Quality of life | up to 3 years

SECONDARY OUTCOMES:
Overall survival | up to 3 years
Toxicity of adjuvant chemotherapy | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Eveline Boucher, MD, Principal Investigator — Centre Eugene Marquis
Locations (37):
- France (37):
  - CHU - Hôpital Nord, Amiens
  - Centre Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Centre hospitalier de la Côte Basque, Bayonne
  - Hôpital Jean Minjoz, Besançon
  - Hôpital Avicenne, Bobigny
  - CHU Brest - Hôpital Morvan, Brest
  - CHU Côte de Nacre, Caen
  - CHU Estaing, Clermont-Ferrand
  - Hôpital Beaujon, Clichy
  - Hôpital Henri Mondor, Créteil
  - Hôpital Bocage, Dijon
  - CHD Vendée, La Roche-sur-Yon
  - Centre Léon Bérard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Saint Joseph, Marseille
  - Hôpital Nord, Marseille
  - Institut Paoli Calmettes, Marseille
  - CHU Timone Adulte, Marseille
  - Centre Hospitalier Saint Eloi, Montpellier
  - Centre René Gauducheau, Nantes
  - Hôpital La Source, Orléans
  - Hôpital Saint Antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Saint Louis, Paris
  - Hôpital de la Pitié Salpétrière, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - CHU de Poitiers, Poitiers
  - Centre Eugene Marquis, Rennes
  - CHU de Rouen - Hôpital Ch. Nicolle, Rouen
  - CHU Sainte-Etienne - Hopital Nord, Saint-Étienne-d'Orthe
  - Centre Paul Strauss, Strasbourg
  - Hôpital de Hautepierre / Hôpital Civil, Strasbourg
  - Hôpital Trousseau, Tours
  - CHU Brabois, Vandouevre Les Nancy
  - Institut Gustave Roussy, Villejuif